CLINICAL TRIAL: NCT05518656
Title: Effects and Mechanisms of Smartphone-Based Stress Management Training on Well-Being in College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20024191
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online emotion regulation training version 1 (Experimental)
  Interventions: Behavioral: Experimental intervention
- Online emotion regulation training version 2 (Active Comparator)
  Interventions: Behavioral: Comparison intervention

INTERVENTIONS:
Behavioral: Experimental intervention — Daily lessons received by email to be completed the same day
  Arms: Online emotion regulation training version 1
Behavioral: Comparison intervention — Daily lessons receive by email to be completed the same day
  Arms: Online emotion regulation training version 2

SUMMARY:
Studying can be a difficult time, and some students can find it challenging to deal with stress. This research project at Virginia Commonwealth University aims to understand how two different online stress management training programs affect students' daily experiences and activities. This research project will help us understand how those training programs help students to improve their emotional well-being.

DETAILED DESCRIPTION:
Participants will be randomly assigned (like the flip of a coin) to one of the two online stress management training programs. For two weeks, participants will receive daily online lessons that will teach you how to deal with stress.

To investigate how this program affects mood, researchers will monitor participant's daily activities and experiences combining brief daily surveys with activity tracking via smartphones. The activities and experiences will be tracked for a week before the training, two weeks of the training, and one week after. Shortly after the training, researchers will also reach out to participants for a phone interview where they will ask about the training experience in more detail. Afterwards, researchers will check in with participants at the end of the semester for one more week of experience and activity tracking.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old;
* Enrollment as a full-time student;
* Studying in-person;
* Reduced emotional well-being;
* Absence of major depressive, generalized anxiety, and panic disorder diagnoses;
* Little or no experience of the intervention;
* Ownership of a smartphone with an OS no older than iPhone 5 or Android 5 and an active data plan.

Exclusion Criteria:

• Diagnosis of major depression, generalized anxiety, and panic disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Change in loneliness | Baseline to the end of the semester, up to 15 weeks
  Loneliness will be measured with the UCLA Loneliness Scale an instrument assessing frequency of felt social disconnection.
Change in social connection | Baseline to the end of the semester, up to 15 weeks
  Connection to others will be measured with the Two-Way Social Support Scale
Change in depression | Baseline to the end of the semester, up to 15 weeks
  Depressive symptoms will be measured using Center for Epidemiologic Studies Depression Scale
Change in anxiety | Baseline to the end of the semester, up to 15 weeks
  Anxiety symptoms will be measured using Beck's Anxiety Inventory
Changes in daily experiences | Baseline to the end of the intervention, 4 weeks
  Smartphone passive sensing will be accomplished through AWARE which will record frequency (but not content) of short message service (SMS) text messaging and calls, location and mobility (to assess out-of-home departures), and nearby Bluetooth addresses (to assess social proximity). A conversation plugin will make surrounding sound inferences (without retaining audio recordings), including presence of other voices.
Changes in daily well-being | Baseline to the end of the intervention, 4 weeks
  Ecological momentary assessment (EMA) will include items to measure mood, loneliness, felt social connection and school belonging, and interactions with others. EMA surveys will be administered through the AWARE app.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Brown, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No